CLINICAL TRIAL: NCT04374045
Title: Testing for Dysautonomia in Patients Hospitalized for SARS-CoV-2 Infection (COVID-19) : COVIDANS Study
Acronym: COVIDANS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH095; 2020-A01082-37 (Other: ANSM)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: SARS-CoV 2
Keywords: COVID-19; SARS-CoV-2; Coronavirus; Dysautonomia
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SARS-CoV-2: patients having a continuous recording of the heart rhythm during their hospitalization
  Interventions: Other: ECG-Holter

INTERVENTIONS:
Other: ECG-Holter — Patient will have a ECG-Holter recording during all their hospitalization.

SUMMARY:
A number of clinical features suggest the possibility of dysautonomia in patients infected with SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2).

At the same time, there is now strong experimental evidence that SARS-CoV-2 can cross the blood-brain barrier, probably via the olfactory nerves, and reach the brain stem, which is located in close proximity.

Damage to the brainstem nuclei could explain the suspected dysautonomic episodes, but also the severity of respiratory distress in infected patients, and the difficulty of ventilatory withdrawal encountered in resuscitation, potentially through damage to the ventilation control and regulation centers located in the brainstem.

The objective of this study is to record the long term variability in heart rate, reflecting autonomic balance, of patients screened positive for SARS-CoV-2 throughout their stay in conventional care units at the Saint-Etienne University Hospital, in order to see whether there is an autonomic imbalance at screening, whether the worsening of the autonomic imbalance precedes the worsening of the clinical condition, and how quickly the expected correction of the autonomic imbalance follows or precedes that of the disease.

DETAILED DESCRIPTION:
In this study, patients will have a continuous recording of their heart rhythm via a holter-ECG throughout their hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* major
* with clinical signs of SARS-CoV-2
* understanding and speaking French fluently to understand the explanations and participate in the study
* who have given their oral consent to participate in the study
* affiliated or entitled to a social security scheme.

Exclusion Criteria:

* with a history of Parkinson's disease, insulin-dependent or non-insulin-dependent diabetes at a dysautonomic stage or chronic alcoholism at a dysautonomic stage
* with atrial fibrillation on the ECG trace taken at the time of their entry.
* refusing to participate in the study
* intubated prior to inclusion in the study
* that are within the exclusion period of another research protocol
* with a history of head injury, neurological pathology with a brain impact, or serious unstable somatic disease
* patient under guardianship.
* pregnancy woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical signs of SARS-CoV-2 (covid-19).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Percentage of dysautonomia patients found within the first 24 hours of hospitalization (%) | Hours: 24
  Dysautonomia will be measured by the LF/HF ratio (sympatho-vagal balance), obtained from a Holter-ECG recording over the first 24 hours of hospitalisation, and compared to normal values given by charts for each age group and sex, making it possible to obtain the percentage of dysautonomic patients.

SECONDARY OUTCOMES:
Analyse the other mathematical indices measuring autonomic balance, obtained by Holter-ECG recording over the first 24 hours and throughout their hospitalisation, in search of possible dysautonomia | up to 5 months
  Measured by the LF/HF ratio (sympathy-vagal balance)
To investigate whether the autonomic balance of patients with CoV-2 SARS correlates with the severity of their clinical condition during their hospital stay. | up to 5 months
  Measured by the LF/HF ratio (sympathy-vagal balance)
To investigate whether the various autonomic parameters recorded are predictive of clinical worsening or improvement, by calculating a prediction threshold for each of the parameters. | up to 5 months
  Measured by the LF/HF ratio (sympathy-vagal balance)

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Hopital nord, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniel M, Charier D, Pereira B, Pachcinski M, Sharshar T, Molliex S. Prognosis value of pupillometry in COVID-19 patients admitted in intensive care unit. Auton Neurosci. 2023 Mar;245:103057. doi: 10.1016/j.autneu.2022.103057. Epub 2022 Dec 17. PMID 36549090